CLINICAL TRIAL: NCT01813812
Title: A Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of DA-6034 and to Demonstrate the Non-inferiority of DA-6034 Compared With Rebamipide in Patients With Acute or Chronic Gastritis
Brief Title: A Study to Evaluate the Efficacy and Safety of DA-6034 and to Demonstrate the Non-inferiority of DA-6034
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA6034_Gas_III (Version 4.3)
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Acute Gastritis; Chronic Gastritis
MeSH Terms: interventions — recoflavone; rebamipide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DA-6034 45mg (Experimental): two tablets (of DA-6034 45mg) are administered for 2 continuous weeks, three times a day.
  Interventions: Drug: DA-6034
- DA-6034 90mg (Experimental): two tablets (of DA-6034 90mg) are administered for 2 continuous weeks, three times a day.
  Interventions: Drug: DA-6034
- Rebamipide 300mg (Active Comparator): two tablets (of Rebamipide 300mg) are administered for 2 continuous weeks, three times a day.
  Interventions: Drug: Rebamipide 300mg

INTERVENTIONS:
Drug: DA-6034
  Arms: DA-6034 45mg; DA-6034 90mg
Drug: Rebamipide 300mg
  Arms: Rebamipide 300mg

SUMMARY:
This is a multicenter, double-blinded, double-dummy, active-controlled, randomized, Phase III clinical trial to evaluate the efficacy and safety of DA-6034 and to demonstrate the non-inferiority of DA-6034 compared with Rebamipide in patients with acute or chronic gastritis. Subjects will receive 45mg, 90mg of DA-6034 and 300mg of Rebamipide, two tablets, three times a day for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute gastritis or chronic gastritis
* 1 or more erosions found in the gastroscope examination
* Age should be: 20≤age≤75

Exclusion Criteria:

* A patient with peptic ulcer and a gastroesophageal reflux disease.
* Received a medication including non-steroid anti-inflammatory drug 2 weeks before the initiation
* Had a surgery regarding gastroesophageal
* A patient with Zollinger-Ellison syndrome
* Had a medical history of a malignant tumor
* A patient who is currently taking anti-thrombotic drugs

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
The number of erosions comparing the before and after the administration. For example, if the number of the erosion is 0, the score is 1 (normal). | 2 weeks
  The scale is classified into 5 steps which are based on the severity of the improvement.
  EX) noticable improvement: 4->1, 3->1, slight improvement: 4->3, 3->2

SECONDARY OUTCOMES:
The number of erosions diagnosed by the gastroscope | 2 weeks
The severity of the digestive symptoms (Scale of 1 to 5) | 2 weeks
  the example of the symptoms are:
  epigastralgia, heartburn, acid reflux, nausea, domperidone

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Chae Jung, M.D., Ph.D., Principal Investigator — Seoul National University Hospital; Soo Heon Park, M.D., Ph.D., Principal Investigator — Catholic University Yeouido St. Mary's Hopspital; Seong Woo Jeon, M.D., Ph.D., Principal Investigator — Kyungpook National University Hospital; Sang Woo Lee, M.D.,Ph.D., Principal Investigator — Korea University Ansan Hospital; Dong Ho Lee, M.D.,Ph.D., Principal Investigator — Seoul National University Bundang Hospital; Kook Lae Lee, M.D., Ph.D., Principal Investigator — SMG-SNU Boramae Medical Center; Ju Yung Cho, M.D., Ph.D., Principal Investigator — Soonchunhyang University Hospital; Ki Myeong Lee, M.D., Ph.D., Principal Investigator — Ajou University School of Medicine; Yongchan Lee, M.D., Ph.D., Principal Investigator — Severance Hospital, Yonsei University; Sang Yong Seol, M.D., Ph.D., Principal Investigator — Inje University; Jeong Seop Moon, M.D., Ph.D., Principal Investigator — Inje University; Jong Sun Rew, M.D., Ph.D., Principal Investigator — Chonnam National University Hospital; Soo Taek Lee, M.D., Ph.D., Principal Investigator — Chonbuk National University Hospital; Chan Kook Park, M.D., Ph.D., Principal Investigator — Chosun University Hospital; Jae Gyu Kim, M.D., Ph.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Sei Jin Youn, M.D., Ph.D., Principal Investigator — Chungbuk National University Hospital; Hak Yang Kim, M.D., Ph.D., Principal Investigator — Hallym University Medical Center; Byung Chul Yoon, M.D., Ph.D., Principal Investigator — Hanyang University; Suck Chei Choi, M.D., Ph.D., Principal Investigator — Wonkwang University Hospital; Ki Nam Shim, M.D., Ph.D., Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea